CLINICAL TRIAL: NCT01010321
Title: Confocal Microscopy of Benign and Malignant Skin Tumors
Status: Suspended | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Aviv Barzilai, Sheba Medical Cener, Dermatology Unit
Other Study IDs: SHEBA-09-7295-AB-CTIL
Record Dates: First submitted 2009-11-02; First posted 2009-11-10 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Skin Cancer
Keywords: skin lesion suspect as BCC or SCC or others
MeSH Terms: conditions — Skin Neoplasms | interventions — Microscopy, Confocal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all study Population: all
  Interventions: Device: confocal microscopy

INTERVENTIONS:
Device: confocal microscopy — non-invasive imaging

SUMMARY:
The investigators speculate that this tool may be used as an alternative and convenient non-invasive diagnostic of skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18
* Skin lesion suspected to either BCC or SCC etc
* Patient was referred for biopsy diagnostic/therapeutic before hand, and regardless of confocal microscope examination, according to the clinical consideration of physician

Exclusion Criteria:

* Pregnant women
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over the age of 18
  - Skin lesion suspected to either BCC,SCC etc
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
efficacy of a confocal microscope as a diagnostic tool | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aviv Barzilai, Dr., Principal Investigator — Sheba Medical Center